CLINICAL TRIAL: NCT02559492
Title: A Platform Study Exploring the Safety, Tolerability, Effect on the Tumor Microenvironment, and Efficacy of INCB Combinations in Advanced Solid Tumors
Brief Title: Itacitinib Combined With INCB024360 and/or Itacitinib Combined With INCB050465 in Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 39110-106
Record Dates: First submitted 2015-09-23; First posted 2015-09-24 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Solid Tumors
MeSH Terms: interventions — itacitinib; INCB039110; epacadostat; parsaclisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A: Itacitinib + epacadostat (Experimental): Group A will utilize an open-label 3+3 dose-escalation design based on observing each dose level for a period of 21 days.
  Interventions: Drug: Itacitinib; Drug: Epacadostat
- Group B: Itacitinib + INCB050465 (Experimental): Group B will utilize an open-label 3+3 dose-escalation design based on observing each dose level for a period of 21 days.
  Interventions: Drug: Itacitinib; Drug: INCB050465

INTERVENTIONS:
Drug: Itacitinib — Itacitinib (INCB039110) tablets will be administered orally once daily in the morning.
  Other Names: INCB039110
  Arms: Group A: Itacitinib + epacadostat
Drug: Epacadostat — Epacadostat tablets will be administered orally, twice daily.
  Arms: Group A: Itacitinib + epacadostat
Drug: Itacitinib — Itacitinib (INCB039110) tablets will be administered orally once daily in the morning.
  Other Names: INCB039110
  Arms: Group B: Itacitinib + INCB050465
Drug: INCB050465 — INCB050465 tablets will be administered orally once daily.
  Arms: Group B: Itacitinib + INCB050465

SUMMARY:
This is an open-label, Phase 1b, platform study in subjects with advanced or metastatic solid tumors. The study will be divided into 3 parts (Part 1a, Part 1b, and Part 2). Part 1a will evaluate a JAK inhibitor with JAK1 selectivity (Itacitinib) in combination with an IDO1 inhibitor (epacadostat; INCB024360; Group A) and Itacitinib in combination with a PI3K-delta inhibitor (INCB050465; Group B) to determine the MTD or PAD and the recommended Part 1b doses for each combination. Once the recommended dose has been identified for each treatment group in Part 1a, subjects with advanced solid tumors will be enrolled into expansion cohorts based upon prior treatment history with a PD-1 pathway-targeted agent (Part 1b). In Part 2, additional expansion cohorts will be enrolled to further evaluate lower doses of itacitinib and INCB050465 in subjects with select tumor types.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18 years or older.
* Willingness to provide written informed consent for the study.
* Part 1a: Subjects with histologically or cytologically confirmed advanced or metastatic solid tumors that have failed prior standard therapy (including subject refusal or intolerance).
* Part 1b: Subjects with endometrial cancer, gastric cancer, head and neck squamous cell carcinoma, melanoma, microsatellite unstable colorectal cancer, non-small cell lung cancer, pancreatic ductal adenocarcinoma, renal cell carcinoma, triple negative breast cancer, or transitional cell carcinoma of the genitourinary tract that have had disease progression after available therapies for metastatic disease that are known to confer clinical benefit, been intolerant to treatment, or refused standard treatment.
* Part 1b: Must have documented confirmed disease progression on a prior programmed cell death-1 (PD-1) pathway targeted agent or must be PD-1 pathway-targeted treatment naïve.
* Part 2: Subjects with HNSCC, NSCLC, pancreatic ductal adenocarcinoma, salivary gland cancer, and transitional cell carcinoma of the genitourinary tract that have had disease progression after available therapies for advanced or metastatic disease that are known to confer clinical benefit, have been intolerant to treatment, or have refused standard treatment.
* Willingness to undergo a pre-treatment and on-treatment tumor biopsy to obtain the specimen.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

Exclusion Criteria:

* Laboratory parameters not within the protocol-defined range.
* Receipt of anticancer medications or investigational drugs within a defined interval before the first administration of study drug.
* Received an immune-suppressive based treatment for any reason within 14 days prior to the first dose of study treatment.
* Has not recovered from toxic effect of prior therapy to < Grade 1.
* Active or inactive autoimmune process.
* Has received a live vaccine within 30 days of planned start of study therapy.
* Active infection requiring systemic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2015-11; Primary Completion 2018-09-10 (Actual); Study Completion 2019-08-18 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Dose Limiting Toxicities (DLTs) | Baseline through 21 days
  Safety and tolerability of the treatment groups.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Every 9 weeks for duration of study participation which is estimated to be 18 months
  Tumor response rates in those subjects with measurable disease.
Progression Free Survival (PFS) | Every 9 weeks for duration of study participation which is estimated to be 18 months
  Progression-free survival, defined as the time from enrollment until the earliest date of disease progression.
Duration of response (DOR) | Every 9 weeks for duration of study participation which is estimated to be 18 months
  Duration of response determined by radiographic disease assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Lance Leopold, MD, Study Director — Incyte Corporation
Locations (11):
- United States (11):
  - Duarte, California
  - Denver, Colorado
  - New Haven, Connecticut
  - Tampa, Florida
  - Chicago, Illinois
  - Rochester, Minnesota
  - Huntersville, North Carolina
  - Nashville, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - Salt Lake City, Utah

REFERENCES:
- [Derived] Naing A, Powderly JD, Nemunaitis JJ, Luke JJ, Mansfield AS, Messersmith WA, Sahebjam S, LoRusso PM, Garrido-Laguna I, Leopold L, Geschwindt R, Ding K, Smith M, Berlin JD. Exploring the safety, effect on the tumor microenvironment, and efficacy of itacitinib in combination with epacadostat or parsaclisib in advanced solid tumors: a phase I study. J Immunother Cancer. 2022 Mar;10(3):e004223. doi: 10.1136/jitc-2021-004223. PMID 35288468